CLINICAL TRIAL: NCT06321575
Title: The Golazo® Peripheral Atherectomy System for a Safe and Effective Atherectomy
Brief Title: The Golazo® Peripheral Atherectomy System for a Safe and Effective Atherectomy (GREAT Trial)
Acronym: GREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avantec Vascular (Industry)
Collaborators: Bright Research Partners (Industry); Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA-CL-5000
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Symptomatic Infrainguinal Peripheral Arterial Disease; Endovascular Intervention
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The investigation is a prospective, multicenter, non-randomized, single-arm, open-label pivotal clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Golazo® Peripheral Atherectomy System (Experimental): Treatment atherectomy of the peripheral vasculature with the Golazo® Peripheral Atherectomy System.
  Interventions: Device: Golazo® Peripheral Atherectomy System (Golazo® Peripheral AS)

INTERVENTIONS:
Device: Golazo® Peripheral Atherectomy System (Golazo® Peripheral AS) — Golazo® Peripheral AS is a sterile, single-use percutaneous device that has two main components: 1) the Golazo® Accustrike atherectomy catheter, and 2) the Golazo® motorized drive unit (MDU) and is intended for use in atherectomy of the peripheral vasculature.

SUMMARY:
The objective of this study is to establish reasonable assurance of safety and effectiveness of the Golazo® Peripheral Atherectomy System when used as indicated in 159 subjects with symptomatic infrainguinal peripheral arterial disease (PAD) in up to 20 investigational sites in the U.S.

DETAILED DESCRIPTION:
The investigation is a prospective, multicenter, non-randomized, single-arm, open-label pivotal clinical study. Subjects will undergo atherectomy treatment with the Golazo® Peripheral Atherectomy System and will then be followed 6-months post-procedure.

ELIGIBILITY:
General inclusion criteria:

1. Age ≥18 years
2. Candidate for atherectomy of the peripheral vasculature in the lower limbs
3. Life expectancy >1 year in the opinion of the investigator
4. Resting ankle brachial index (ABI) ≤0.90, or ≤0.75 after exercise. Subjects with non-compressible arteries shall have a toe brachial index (TBI) assessment.
5. Target limb Rutherford clinical classification category 3 to 5
6. Suitable candidate for angiography and endovascular intervention in the opinion of the investigator
7. Willing and able to comply with the protocol-specified procedures and assessments
8. Informed consent granted

   Angiographic inclusion criteria:
9. Target lesion(s) defined as stenosis ≥70% by angiographic visual estimation
10. Total treated lesion length ≤20 cm by angiographic visual estimation
11. Target reference vessel diameter (RVD) ≥2.0 mm and ≤4.5 mm by angiographic visual estimation
12. Target limb will have a minimum of one patent (less than 50% stenosis) below the knee (BTK) vessel crossing the ankle, distal to any target lesion, providing perfusion to the foot at baseline

General exclusion criteria:

1. Active infection in the target limb
2. History of an endovascular procedure or open vascular surgery on the target limb within the last 30 days
3. Planned surgical or interventional procedure within 30 days after the index procedure
4. Lesion in the contralateral limb requiring intervention during the index procedure or within next 30 days
5. Critical limb ischemia (CLI) with Rutherford clinical classification category 6
6. Significant acute or chronic kidney disease with a GFR <30 and/or requiring dialysis
7. Acute myocardial infarction (non-ST-elevation myocardial infarction or ST-segment elevation myocardial infarction) or other uncontrolled comorbidity in the opinion of the investigator
8. Myocardial infarction (MI) or stroke within two months of baseline evaluation
9. Pregnant or lactating
10. Subject is participating in another clinical investigation of a device, drug, or procedure that has not completed the study treatment or that clinically interferes with the endpoints of this study (post-approval registries are allowed as long as the investigator determines there is no clinical interference with study endpoints)
11. Contraindication to antiplatelet, anticoagulant, or thrombolytic therapy
12. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count <125,000/microliter, known coagulopathy, or international normalized ratio (INR) >1.5
13. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately medicated
14. History of heparin-induced thrombocytopenia (HIT)
15. Any thrombolytic therapy within two weeks of enrollment
16. Target lesion(s) within a native vessel graft or synthetic graft
17. Significant stenosis or occlusion of inflow not successfully treated before the index procedure
18. Any evidence or history of intracranial or gastrointestinal bleeding or intracranial aneurysm
19. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults)
20. One or more of the following complications of the foot:

    1. Osteomyelitis that extends to the metatarsal bones.
    2. Gangrene involving the plantar skin of the forefoot, midfoot or heel
    3. Deep ulcer or large shallow ulcer (>3cm) involving the plantar skin of the forefoot, midfoot, or heel
    4. Any heel ulcer with/without calcaneal involvement
    5. Any wound with calcaneal bone involvement
    6. Wounds that are deemed to be neuropathic or non-ischemic in nature
    7. Wounds that require flap coverage or complete wound management for large soft tissue defect
21. Congestive heart failure with a NYHA functional classification of III or higher

    Angiographic exclusion criteria:
22. More than 2 lesions to be treated with the investigational device; lesions located within 3 mm may be considered a single tandem lesion
23. Clinical/angiographic complication (other than non-flow limiting dissections) attributed to a currently marketed device prior to introduction of the investigational device
24. In-stent restenosis within the target lesion(s)
25. Potentially unstable or flow-limiting dissection, type C or greater
26. Clinical/angiographic evidence of distal embolization
27. Inability to cross the proximal lesion vessel lumen with a guidewire (not subintimal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events (MAE) | Index procedure through 30-day follow-up
  MAE is defined as:
  * Clinically-driven target lesion revascularization (CD-TLR)
  * Cardiovascular-related deaths
  * Unplanned major target limb amputation (above the ankle)
  * Perforations or dissections grade C or greater in the target vessel that require intervention
  * Symptomatic distal emboli requiring intervention
  * Pseudoaneurysm requiring intervention
Technical success | During surgery/procedure
  Defined as the percent of target lesions that have a residual diameter stenosis ≤50% after atherectomy with the Golazo Peripheral AS and prior to adjunctive therapy

SECONDARY OUTCOMES:
Change in % stenosis in target lesion after treatment with Golazo Peripheral AS | During surgery/procedure
  Determined after atherectomy and prior to other adjunctive therapies
Procedural Success Rate | End of surgery/procedure
  Defined as the proportion of the target lesion in which the final stenosis is ≤30% after treatment with atherectomy and any other adjunctive therapy
Clinical Success Rate | 30-day and 6-month follow-up
  Defined as the proportion of subjects who have procedural success in all target lesions with at least one grade of improvement in the Rutherford clinical classification
Rates of all adverse events classified as MAEs | 30-day and 6-month follow-up
  As adjudicated by the CEC and presented by seriousness and causality (procedure and device relatedness)
Incidence of minor target limb amputation | 30-day and 6-month follow-up
  As adjudicated by the CEC
Incidence of myocardial infarction | 30-day and 6-month follow-up
  As adjudicated by the CEC
Incidence of target vessel revascularization (TVR) in the target limb | 30-day and 6-month follow-up
  As adjudicated by the CEC
Incidence of angiographic procedural distal embolization in the target limb | During surgery/procedure
  As reported by the angiographic core laboratory
Time to primary patency of the target lesion(s) | 6 months
  Primary patency is the interval from the time of the index procedure until the time of any intervention designed to maintain or reestablish patency of the target vessels, the time significant stenosis or total occlusion is confirmed, or the time of measurement of patency. Determined by duplex ultrasound/doppler (DUS) or angiography.
Time to assisted primary patency of the target lesion(s) | 6 months
  Assisted primary patency is the interval from the time of the index procedure until the time significant stenosis is confirmed, including interventions designed to maintain patency of a vessel with significant stenosis, the time total occlusion is confirmed, or the time of measurement of patency. Determined by duplex ultrasound/doppler (DUS) or angiography.
Time to secondary patency of the target lesion(s) | 6 months
  Secondary patency is the interval from the time of the index procedure until the time total occlusion is confirmed in a target vessel, including interventions designed to reestablish patency in a total occluded vessel, or the time of measurement of patency. Determined by duplex ultrasound/doppler (DUS) or angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Finn, MD, Principal Investigator — Cardiovascular Institute of the South; Craig Walker, MD, Principal Investigator — Cardiovascular Institute of the South
Locations (20):
- United States (20):
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Pulse Cardiovascular Institute, Scottsdale, Arizona
  - Merced Vascular, Merced, California
  - Palm Vascular Center, Fort Lauderdale, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Radiology and Imaging Specialists of Lakeland, Lakeland, Florida
  - Amavita Research Services, Miami, Florida
  - Cardiovascular Consultants of South Georgia, Thomasville, Georgia
  - Pacific Vascular Institute, ‘Aiea, Hawaii
  - Baton Rouge General Hospital, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South - Houma, Houma, Louisiana
  - Cardiovascular Institute of the South - Lafayette, Lafayette, Louisiana
  - Vascular Breakthroughs, Plymouth, Massachusetts
  - Advanced Heart and Vascular Institute, Flemington, New Jersey
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Nextstage Clinical Research - Beaumont, Beaumont, Texas
  - Hope Vascular & Podiatry, Houston, Texas
  - Nextstage Clinical Research - Waco, Waco, Texas
  - Bellin Health, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No